CLINICAL TRIAL: NCT02343731
Title: Dogs as Probiotics to Enhance the Health and Emotional Well-Being of Elderly Adults
Brief Title: Dogs as Probiotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ole Thienhaus, Director, Department of Psychiatry; College of Medicine, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pending NCT02343731
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Health of the Human Microbiome
Keywords: microbiome; hygiene hypothesis; human-animal interaction; microbiota; connections between human-canine microbiome
MeSH Terms: conditions — Human-Animal Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dog Introduction (Experimental): Participants will receive a dog from the Humane Society of Southern Arizona's (HSSA) foster care program to live with them for three months.
  Interventions: Other: Introduction of a dog into the home

INTERVENTIONS:
Other: Introduction of a dog into the home — Participants will foster dogs from the HSSA for three months while they are in the study.

SUMMARY:
Studies show that family members share as much or more of the composition of their microbiota (the trillions of micro-organisms in our guts) with their dogs as they do with each other (Song et. al. 2013). This shows that the introduction of dogs into home environments has a profound impact on the human microbiota. Additionally, many studies show that children raised with dogs are less likely than others to develop a range of immune-mediated disorders, including asthma and allergies (Ownby, Johnson, and Peterson 2002; Almqvist et al. 2003; Havstad et al. 2011). This suggests that dogs can serve as probiotics for children by appropriately training their immune systems not to produce inflammation in response to harmless stimuli. What is not known, however, is whether the same is true for elderly populations and dogs. Thus, this study seeks to explore whether dogs might also improve the physical and mental health of elderly adults by improving the structure and function of their microbiota. The investigators propose a pilot/proof of concept study to investigate whether dogs might improve the physical and mental health of elderly adults via changing (improving) the structure and function of their microbiota (gut flora). The investigators propose a pre-post study design that among 20 elderly individuals (aged 50 and older) to investigate the probiotic effect that dogs might have on these individuals. The investigators are particularly interested to know whether introducing a dog into a home where one has not lived in the recent past increases the "positive" microorganisms in the guts of the humans living with them. The investigators will also measure the changes in markers of inflammation (from blood samples) as well as the changes in self-reported scores of depression, frailty, physical activity, and general health and well-being mobility among human participants. In order to assess any effects in the animal study participants, the investigators will also collect and analyze fecal and blood samples as well as conduct home visits to observe canine and human interactions and bonding and conduct assessments of canine well-being using questionnaires/observational techniques that have been validated for these purposes in other studies. Additionally, the investigators will assess the interactions between of the participants with the dog and how having a dog in the home may influence an individual's relationship with the dog and his/her thoughts about the microbiota, human and canine health and human-animal interactions through monthly semi-structured interviews.

The investigators have previously received IACUC approval for this study, approval number 14-537.

DETAILED DESCRIPTION:
One of the most amazing scientific discoveries of the last decade has been the important roles that the trillions of micro-organisms in our guts (called the "microbiota") play in promoting good physical health and emotional well-being. Unfortunately, many aspects of the modern world conspire to alter the composition and function of the gut microbiota in ways that damage health, especially in the elderly where strong correlations have been seen between microbiota composition and frailty. Work from our research group and others suggests that one very important factor that damages the microbiota in the modern world is our separation from many micro-organisms with which the investigators co-evolved and which have the ability to lower the types of chronic inflammation that are ubiquitous in the modern world and that contribute to the development of most of our most pressing health issues, from diabetes and heart disease to depression and dementia (Huang et al., 2013; Mayer et al, 2014; Naseribafrouei, 2013). While much has been written about the positive psycho-social impacts that animal-human relationships have on human psychological health (Allen et al, 1991; Allen et al.; 2002; Collins et al, 2006; Kwong & Bartholomew, 2011; Kurdek, 2008; Wells, 2007), less is known about the direct physical effects that animals have on human health. What is known, however, is largely related to animals' effects on stress reduction (Allen et al, 1991; Allen et al., 2002) anxiety (Foster & McVey Neufeld, 2013), mood (Collins et al, 2006) and cardiovascular disease (Allen et al., 2002) What has been largely unexplored, however, is the mechanism by which these interactions and positive impacts on human health are taking place. Thus, working with colleagues who are world leaders in studying links between the microbiota and health, the investigators propose to conduct a study designed to explore the potential of dogs to serve as "probiotic delivery systems" to enhance the physical health and cognitive and emotional functioning of at-risk elderly persons.

The rationale for this novel approach to enhancing health and well-being in the elderly comes from several lines of evidence. First, one recent study shows that family members share as much or more of the composition of their microbiota with their dogs as they do with each other (Song et al. 2013). This shows that the introduction of dogs into home environments has a profound impact on the human microbiota. Second, many studies show that children raised with dogs are less likely than others to develop a range of immune-mediated disorders, including asthma and allergies (Ownby et al. 2002; Almqvist et al. 2003; Havstad et al. 2011). This suggests that dogs can serve as probiotics for children by appropriately training their immune systems not to produce inflammation in response to harmless stimuli. Thus, what is not known, and what this study is designed to explore, is whether dogs might also improve the physical and mental health of elderly adults by improving the structure and function of their microbiota. This is a proof of concept / pilot study. Should results from this study suggest that there is indeed a positive benefit/relationship to canine companionship to the microbiota of elderly human companions, the investigators plan to implement a larger, full-scale clinical trial to investigate this phenomenon.

Hypothesis: The investigators hypothesize that the introduction of a canine companion into the home of an elderly individual (defined as aged 50 and older) will result in an increase in protective or 'positive' gut micro-organisms and that this increase will correspond with improved immune functioning in the elderly human study participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or females aged 50 - 80.
* In general good health (mobile and able to care for a dog).
* Have not taken antibiotics in the last six months.
* Have not had a dog in the home for the past six months.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* Able to communicate in English with study personnel.
* Willing to commit to fostering a dog for at least three months with the understanding that at the end of the three months, they can keep the dog if they so desire.

Exclusion Criteria:

* Individuals who are currently on any antibiotic therapy. Participants who are on an antibiotic therapy will be allowed to participate in the study after a six month washout period.
* Unwilling to have a dog in the home for at least three months of time.
* Any of the following diagnoses, as identified by the intake evaluation conducted or study assessments:

  o History of any of the following mental illnesses: schizophrenia, bipolar I disorder, drug or alcohol abuse active within 6 months of study entry. Determination of these criteria will be by self-report at screening interview
* Subject has a medical condition or disorder that:

  * Is unstable and clinically significant, or:
  * Specifically impact immune functioning of the GI tract including Crohn's disease and ulcerative colitis
  * Require either chronic or periodic antibiotic treatment
  * Could interfere with the accurate assessment of safety or efficacy of the clinical assessments, including:
* Individuals with any:

  o Current participation in any clinical trial that might impact results of this one, which includes participation in another clinical trial where any experimental drugs are being taken as well as studies / drug trials with agents that might affect mood and or the gastrointestinal tract.
* Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.
* Any clinically significant autoimmune disease (compensated hypothyroidism allowed)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Increase in positive microbiota in humans | Seven days prior to the intervention, Day 0, Day 30, Day 60 and Day 90
  To examine the degree to which the positive microbiota increase in human study participants' guts from baseline to three months. We will do this by collecting the human participants' saliva, skin and feces.
Correlation between positive microbiota changes and immune function changes | Seven days prior to the intervention, Day 0, Day 30, Day 60 and Day 90
  To examine the correlations between positive microbiota changes in the human gut after introduction of a canine companion with any changes in immune and related molecules that have been linked to emotional well-being. We will do this by collecting blood from the human participants.

SECONDARY OUTCOMES:
Change in human physical activity over time | Seven days prior to the intervention, Day 0, Days 23-30, Days 53-60 and Days 83-90
  The study participant will wear a non-invasive Actigraph GT3X+ device which clips to the waistbelt for 7 consecutive days at 4 time points in the study. The accelerometer is small (1.5x2 inches) and will be clipped to the waistband/belt.
Change in dog physical activity over time | Seven days prior to the intervention, Day 0, Days 23-30, Days 53-60 and Days 83-90
  Whistle monitors are pet activity monitors that dogs can wear around their necks, attached to their dog collars. Whistle monitors come with a built-in accelerometer that senses the animal's movement. The accelerometer measures steps taken, distance walked, and overall activity duration and intensity every 30 seconds.
Change in heart rate variability over time | Day 0, Day 30, Day 60 and Day 90
  Heart Rate Variability (HRV) will be assessed over time to see if having a dog significantly impacts HRV. HRV will be assessed during the period of SCL collection and will be calculated using both time and frequency domain methodologies.
Change in frailty score over time | Day 0, Day 30, Day 60 and Day 90
  The Fried Frailty test will be administered and changes in participants overall schedule will be assessed and compared over time.
Change in body fat composition over time | Day 0, Day 30, Day 60 and Day 90
Change in Score on the Q-LESQ-SF (Quality of Life Enjoyment and Satisfaction Questionnaire -Short form) | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores between baseline and subsequent assessments will be assessed to determine the effect of dog ownership on self-reported quality of life.
Change in score on the WHO-5 | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores between baseline and subsequent visits on the WHO-5, to assess the effect of dog ownership on current well being.
Change in depression scores over time [Inventory of Depressive Symptomatology-Self Report (IDS-SR)] | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores between baseline and subsequent assessments will be assessed to determine the effect of dog ownership on any depression symptoms.
Change in scores over time Short Form-36 | Day 0, Day 30, Day 60 and Day 90
  Percent change in the SF-36, a standard health questionnaire that assesses dog ownerships effect on overall physical health and emotional well-being.
Change in scores over time on the UCLA Loneliness Scale | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores on the UCLA Loneliness Scale to assess the effect of dog ownership on loneliness.
Change in scores over time on the Mini-Cognition Test | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores on the Mini-Cognition Test to assess the effect of dog ownership on cognition over time.
Change is scores over time on the International Physical Activity Questionnaire (IPAQ) | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores on the Physical Activity Questionnaire (IPAQ) is a short standard questionnaire to assess the effect of dog ownership on physical activity.
Change in scores over time on the Dogs and Physical Activity Tool (DAPA) | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores on the DAPA to assess effect of dog ownership on dog physical activity.
Change in scores over time on the Dog Quality of Life Scale | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores on the Dog Quality of Life Scale to assess the effect of dog ownership on a dog's quality of life.
Change in scores over time on the Lexington Human Animal Bond (HAB) | Day 0, Day 30, Day 60 and Day 90
  Percent change in scores on the HAB measure to assess how the human animal bond changes over the study period.
Interviews | Day 0, Day 30, Day 60 and Day 90
  The topics to be covered in the interview will include a discussion of previous dog/animal ownership, thoughts and feelings on the animal-human bond, understandings of the microbiota, animal-human microbiota connections and intersections between animals, humans and scientific understandings of the body and medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Study Director — University of Arizona, Department of Psychiatry, College of Medicine; Ole Thienhaus, MD, Principal Investigator — University of Arizona, Department of Psychiatry, College of Medicine
Locations (1):
- University of Arizona, Tucson, Arizona, United States